CLINICAL TRIAL: NCT00664898
Title: An Open-Label, Phase Ib, Dose-Escalation Study of the Safety and Pharmacology of the Anti-CD40 Monoclonal Antibody SGN-40 Administered in Combination With Bortezomib (Velcade®, PS-341) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of the Safety and Pharmacology of SGN-40 Administered in Combination With Bortezomib in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACF4375g
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Multiple Myeloma
Keywords: anti-CD40; Myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; dacetuzumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bortezomib; Drug: SGN-40

INTERVENTIONS:
Drug: bortezomib — Escalating intravenous repeating dose
Drug: SGN-40 — Escalating intravenous repeating dose

SUMMARY:
This is an open-label, multicenter, Phase Ib study to be conducted at approximately eight sites in Europe and the U.S. designed to evaluate the safety, pharmacokinetics, and activity of SGN-40 when combined with bortezomib in patients with multiple myeloma that is relapsed or refractory after at least one prior systemic treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Documented pathologic diagnosis of multiple myeloma that has relapsed or failed to respond after treatment with at least one prior systemic therapy (other than corticosteroid monotherapy)
* Measurable disease
* At least one prior systemic therapy other than single-agent corticosteroids
* European Union patients must have had prior bone marrow transplant (autologous) or be ineligible for transplant
* If previously received bortezomib, demonstration of clinical response of any duration or stable disease with progression-free interval of ≥ 6 months from the start of that therapy
* If previously received bortezomib, must have recovered from bortezomib-related toxicities and must have a peripheral neuropathy score of Grade ≤ 1, according to the NCI CTCAE v3.0
* If applicable, completion of autologous transplant ≥ 12 weeks prior to Day 1
* Discontinuation of previous anticancer or investigational therapy for ≥ 21 days prior to treatment, or ≥ 90 days prior to treatment for previous monoclonal antibody administration

Exclusion Criteria:

* Prior allogeneic bone marrow transplant
* Other invasive malignancies within 3 years prior to Day 1 except for adequately treated basal cell or squamous cell skin cancer; carcinoma in situ of the cervix, breast, or prostate; or other cancer of which the patient has been disease-free for ≥ 3 years
* Prior anaphylactic reaction to human immunoglobulin administration
* Symptomatic hyperviscosity syndrome
* Active infection requiring parenteral antibiotics within 14 days of Day 1
* Major surgical procedure or significant traumatic injury within 28 days prior to Day 1, or anticipation of need for major surgical procedure during the course of the study
* Clinically significant cardiac dysfunction or other significant organ dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-05; Primary Completion 2010-04-08 (Actual); Study Completion 2010-04-08 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of SGN-40 when combined with bortezomib | Length of study

SECONDARY OUTCOMES:
Determine safety, pharmacokinetics, and clinical response rate for combination therapy with SGN-40 and bortezomib | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Skettino, M.D., Study Director — Genentech, Inc.